CLINICAL TRIAL: NCT03341182
Title: The Effects of Use of Mirror Image on Radiation Exposure During Fluoroscopically Guided Transforaminal Epidural Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 4-2017-0801
Record Dates: First submitted 2017-10-25; First posted 2017-11-14 (Actual); Last update posted 2019-01-22 (Actual); Status verified 2019-01

CONDITIONS: Lumbar Radiculopathy Due to Spinal Nerve Compression
Keywords: epidural steroid injection; radiation exposure; mirror

STUDY DESIGN:
Intervention Model Description: normal method group (group A) mirror use group (group B)
Who Masked: Participant, Investigator
Masking Description: 1. The subjects were randomly assigned to normal method group (group A) and mirror use group (group B), and the assigned results are unknown.
  2. The Outcomes Assessor is not related to the study, and does not know its contents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- normal method group (group A) (Active Comparator): A mirror is not used in tunnel view technique (conventional manner)
  Interventions: Procedure: conventional manner
- mirror use group (group B) (Experimental): A mirror is used in tunnel view technique
  Interventions: Procedure: Fluoroscopically Guided Lumbar Transforaminal Epidural Injections

INTERVENTIONS:
Procedure: Fluoroscopically Guided Lumbar Transforaminal Epidural Injections — Lay the subject down on the stomach and hold the pillow on the stomach. The skin of the injection area is sterilized by aseptic method and covered with aseptic pouch. After confirming the level of he vertebrae around the C-arm and aligning the anteroposterior view of the endplate of the vertebral body, rotate the C-arm 20~30 degrees diagonally in the direction to be performed. After confirming the best Scotty dog view, confirm the final target point at 6 o'clock directly below the pedicle. At this position, the skin point is marked on the skin. And then both groups proceed in parallel with the beam direction of the transducer with the tunnel view technique until the needle reaches the back of the vertebral body at the level of the spinal nerve roots. At this time group A uses a mirror and group B dose not. The final reach of the target point (ideal depth) is confirmed through the anterior and posterior views and lateral views.
  Arms: mirror use group (group B)
Procedure: conventional manner — A portable mirror is located at the side of surgical table and used in this procedure.
  Arms: normal method group (group A)

SUMMARY:
Lumbar Transforaminal Epidural Injection is helpful for the treatment of lumbosacral radicular pain.

Tunnel view technique is the basis of X-ray assisted intervention. In this technique, it is necessary to handle the block needle in order to adjust the direction of needle to the tunnel view toward target. If a mirror is used during needle handling, overall procedure time and radiation exposure can be reduced.

DETAILED DESCRIPTION:
1. A planned Fluoroscopically Guided Lumbar Transforaminal Epidural Injection should be performed after receiving the informed consent of the patient.
2. This study is single-blind because it is not possible to blind the practitioner performing the injection.
3. Subjects were randomly assigned to the normal method group (group A) and the mirror use group (group B) by a random random number table, and the possibilities for belonging to any group were all the same and can not be artificially controlled by researchers.
4. After the procedure, a resident who does not know of this study records the radiation exposure time displayed on the monitor and the overall procedure time

ELIGIBILITY:
Inclusion Criteria:

1. Magnetic resonance imaging (MRI) and clinical manifestations of adult men and women over 20 years of age are eligible for radiculopathy due to back nerve root compression and subject to fluoroscopically guided lumbar transforaminal epidural Injection at the suspected spinal nerveroots level.

Exclusion Criteria:

1. Blood clotting disorder
2. Infection around the site
3. Contrast agent allergy
4. Uncontrolled cardiovascular, cerebrovascular, kidney disease
5. Past history of spinal surgery (ex, spinal fusion)
6. If can not block due to Non-cooperation with subjects (ex, if you can not take the stomach)
7. Patients taking narcotic analgesics

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-12-21 (Actual); Primary Completion 2018-08-21 (Actual); Study Completion 2018-08-21 (Actual)

PRIMARY OUTCOMES:
radiation exposure time(second) | Immediately after the procedure
  In both groups, overall procedure time recorded on the monitor is recorded after the procedure is over.

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Anesthesiology and Pain Medicine, Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No